CLINICAL TRIAL: NCT01370057
Title: The Use of TLSOs in the Treatment of Adolescent Idiopathic Scoliosis: A Prospective, Randomized Controlled Study
Brief Title: The Use of Thoraco-lumbo-sacral Orthoses (TLSOs) in the Treatment of Adolescent Idiopathic Scoliosis (AIS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure of Subject Recruitment
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHENG Chun-yiu Jack, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRAIST HK PROTOCOL VER1
Record Dates: First submitted 2011-05-20; First posted 2011-06-09 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Scoliosis; AIS; Brace; TLSO
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Treatment with bracing
  Interventions: Device: Thoraco-lumbo-sacral Orthosis
- Control Group (No Intervention): Watchful waiting without bracing

INTERVENTIONS:
Device: Thoraco-lumbo-sacral Orthosis — Treatment with Thoraco-lumbo-sacral Orthosis for Adolescent Idiopathic Scoliosis
  Other Names: The Thoraco-lumbo-sacral Orthosis is fabricated at Prosthetic & Orthotic Department at our research facility(Prince of Wales Hospital, Hong Kong SAR, China)
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to compare the risk of curve progression in Adolescent Idiopathic Scoliosis for subjects treated with bracing as compared to those without bracing.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of AIS
* Age ≥10, ≤15 years old
* Risser 0, 1 or 2
* Primary Cobb angle between 20 and 40 degrees (inclusive)
* Apex (of at least one of the primary curves) caudal to T7
* Pre-menarchal OR post-menarchal by ≤1 year
* Physical and mental ability to adhere to bracing protocol

Exclusion Criteria:

* Diagnosis of other musculoskeletal or developmental illnesses possibly responsible for the curvature
* A history of previous surgical or orthotic treatment
* Inability to read and understand Chinese

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2011-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Curve progression | Till cessation of growth or progression of curve severity to 50 degrees or more, patient will be followed once every 6 months, an average follow up of 3 years is expected
  Curve progression to Cobb angle of 50 degrees or more

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, China